CLINICAL TRIAL: NCT04754607
Title: Effects of Low-Level Laser Therapy on Oxidative Stress Levels and Quality of Life in Patients With Hashimoto Thyroiditis
Brief Title: Effects of Low-Level Laser Therapy on Oxidative Stress Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, sumeyye tunc, MSc, Physiotherapist, Lecturer, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMU-FTR-ST-01
Record Dates: First submitted 2021-02-12; First posted 2021-02-15 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Hashimoto Thyroiditis; Autoimmune Thyroiditis; Thyroiditis; Thyroid Diseases; Autoimmune Diseases
Keywords: Hashimoto Thyroiditis; Oxidative Stress; Low-Level Laser Therapy; Quality of Life; Autoimmune Thyroiditis; Thyroid Hormones; Photobiomodulation Therapy
MeSH Terms: conditions — Hashimoto Disease; Thyroiditis, Autoimmune; Thyroiditis; Thyroid Diseases; Autoimmune Diseases | interventions — Low-Level Light Therapy; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Level Laser Therapy Group (Active Comparator): Low Level Laser Therapy (LLLT): Low-level laser therapy will be applied to the cases in addition to LT4 hormone replacement therapy.
  LLLT group will be treated using a continuous wave GaAIAs type diode laser (Intelect® Mobile Laser, Model No: 2779, Production Year: 2016; Chattanooga Group) device in the treatment area of 0.07 cm2. Continuous mode at 850 nm wavelength, 100 mW output power,1.43 W/cm2 power density and 28.57 J / cm2 energy density will be used.
  Interventions: Other: Low Level Laser Therapy
- Sham Group (Sham Comparator): Probes were placed in the sham laser group in a similar way as in the treatment group.
  Interventions: Other: Sham

INTERVENTIONS:
Other: Low Level Laser Therapy — Eight target points (superior, mediolateral, inferior border of the right and left thyroid lobes, right and left sides of the isthmus) will be marked with a surgical pen by determining the thyroid borders on the skin by thyroid ultrasonography by the specialist physician. Low-level laser (28.57 J / cm2) fixed applications will be made on the thyroid gland, approximately 1 cm from each other. In practice, the patient's neck will be maintained in the extension position. Each application will last 20 seconds and the radiant energy will be 2 J, the tip of the laser will be kept in contact with the skin and upright. Duration of treatment is 6 sessions 2 days a week. The cumulative dose will be 96 J.
  Arms: Low Level Laser Therapy Group
Other: Sham — Probes were placed in the sham laser group in a similar way as in the treatment group. The screen of the laser device was active; however, the energy was set as 0 J and the power as 0 mW , respectively,and the same operations were also performed.
  Arms: Sham Group

SUMMARY:
Hashimoto's thyroiditis (HT) is the most commonly observed inflammatory and autoimmune disease of the thyroid gland. Recent evidence has suggested that low-level laser therapy (LLLT) can improve thyroid function and reduce levels of thyroid peroxidase antibodies (TPOAb) in patients with hypothyroidism caused by chronic autoimmune thyroiditis. In the literature, data examining the effects of LLLT on oxidative stress level and quality of life in patients with HT is limited. The aim of the study is to examine the effects of LT4 treatment combined with LLLT on thyroid autoimmunity, oxidative stress and quality of life in patients with Hashimoto's diagnosis.

DETAILED DESCRIPTION:
Hashimoto's thyroiditis (HT) is the most commonly observed inflammatory and autoimmune disease of the thyroid gland. HT is the main cause of spontaneous hypothyroidism in adults. Symptoms of hypothyroidism may develop within a few years in patients with initial euthyroidism. Many genetic and environmental factors play a role in the pathogenesis of the disease, including iodine exposure, drugs, chemicals, toxins, infections and smoking. In recent years, the relationship between oxidative stress level and thyroid autoantibodies in HT has attracted increasing attention of researchers. In the studies, it has been reported that oxidative stress levels may increase due to chronic inflammation, insufficient thyroid hormone levels, excessive autoimmune response and excessive iodine intake. OS occurs as a result of an imbalance between free radical production and antioxidant defense mechanisms. Data from clinical studies clearly show that the balance between oxidants and antioxidants shifts towards the oxidative side in patients with autoimmune thyroiditis, suggesting that oxidative stress may be a key event in the pathophysiology of the disease, independent of thyroid function. Gerenova et al. divided patients with a diagnosis of HT into three subgroups according to thyroid function (group 1-euthyroid, group 2-hypothyroid, and group 3-Levothyroxin treated patients) and pointed out cellular antioxidative deficiency in all stages of the disease. Standard treatment in patients with HT is lifelong levothyroxine (LT4) treatment, which adjusts the dose to reach normal circulating thyrotropin (TSH) levels. Studies have found persistent fatigue, psychological and general well-being, and impairments in cognitive function in patients with HT despite LT4 replacement therapy. Gomez et al. compared 152 hypothyroid women treated with levothyroxine and 238 women without hypothyroidism disorder. Female patients with hypothyroidism, despite being euthyroid, showed worse quality of life than the control group. It was emphasized that the quality of life of women with hypothyroidism should be evaluated and further research should be conducted. Recent evidence has suggested that low-level laser therapy (LLLT) can improve thyroid function and reduce levels of thyroid peroxidase antibodies (TPOAb) in patients with hypothyroidism caused by chronic autoimmune thyroiditis. LLLT is a non-invasive, painless, low-risk and low-cost method that uses the interaction of light with molecular structures to support anti-inflammatory effects and regeneration of biological tissues. In the literature, data examining the effects of LLLT on oxidative stress level and quality of life in patients with HT is limited. As far as we know, it will be the first study examining the effect of LLLT on oxidative stress and quality of life in cases diagnosed with HT. The planned research is trying to improve and expand the existing literature on LLLT in cases with HT and to contribute to the treatment protocol in order to reduce the negative consequences that may be experienced in this group of patients now and in the future. These statements show the originality of the study. Purpose: The aim of the study is to examine the effects of LT4 treatment combined with LLLT on thyroid autoimmunity, oxidative stress and quality of life in patients with Hashimoto's diagnosis.

ELIGIBILITY:
Inclusion Criteria:

Cases between the ages of 18-65 who applied to the Kosuyolu Istanbul Medipol Hospital Endocrinology and Metabolic Diseases Clinic between 2020-2021 and diagnosed as "Hashimoto Thyroiditis" by a specialist physician will be included in the study.

Exclusion Criteria:

* Acute infection
* Use of immunosuppressants, immunostimulants and drugs that interfere with the production, transport, and metabolism of thyroid hormones
* Thyroid nodules
* Tracheal stenosis
* Serious illness
* History of exposure to ionizing radiation and/or neoplasia in the cervical region
* Malignancy and a history of thyroid surgery
* Hypothyrodism caused by postpartum thyroiditis
* Pregnancy and breastfeeding period
* Identification and diagnosis of the cases with neurological and psychiatric disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Oxidative Stress Levels | 3 months
  Biochemical parameters will be taken from the patient file routinely requested by the physician. For routine or whole blood analysis, leftover serum samples will be collected from the blood taken after fasting for 10-12 hours and the separated serum samples will be kept in a -80 °C refrigerator until the analysis day. The analysis of the collected samples will be examined in the Biochemistry Laboratory of Istanbul Medipol University. Oxidative Stress Index (OSI) will be calculated by measuring Total Oxidant Level (TOS) and Total Antioxidant Levels (TAS).
Malondialdehyde (MDA) | 3 months
  For routine or whole blood analysis, leftover serum samples will be collected from the blood taken after fasting for 10-12 hours and the separated serum samples will be kept in a -80 °C refrigerator until the analysis day. The analysis of the collected samples will be examined in the Biochemistry Laboratory of Istanbul Medipol University. Oxidative stress biomarkers will be examined.
Nitric oxide (NO) | 3 months
  For routine or whole blood analysis, leftover serum samples will be collected from the blood taken after fasting for 10-12 hours and the separated serum samples will be kept in a -80 °C refrigerator until the analysis day. The analysis of the collected samples will be examined in the Biochemistry Laboratory of Istanbul Medipol University. Oxidative stress biomarkers will be examined.
Superoxide dismutase (SOD) | 3 months
  For routine or whole blood analysis, leftover serum samples will be collected from the blood taken after fasting for 10-12 hours and the separated serum samples will be kept in a -80 °C refrigerator until the analysis day. The analysis of the collected samples will be examined in the Biochemistry Laboratory of Istanbul Medipol University. Oxidative stress biomarkers will be examined.
Catalase (CAT) | 3 months
  For routine or whole blood analysis, leftover serum samples will be collected from the blood taken after fasting for 10-12 hours and the separated serum samples will be kept in a -80 °C refrigerator until the analysis day. The analysis of the collected samples will be examined in the Biochemistry Laboratory of Istanbul Medipol University. Oxidative stress biomarkers will be examined.
Glutathione (GSH) | 3 months
  For routine or whole blood analysis, leftover serum samples will be collected from the blood taken after fasting for 10-12 hours and the separated serum samples will be kept in a -80 °C refrigerator until the analysis day. The analysis of the collected samples will be examined in the Biochemistry Laboratory of Istanbul Medipol University. Oxidative stress biomarkers will be examined.

SECONDARY OUTCOMES:
Quality of life (QOL) | 3 months
  Short Form-36 questionnaire: The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.

CONTACTS AND LOCATIONS:
Overall Officials: Şükriye Leyla ALTUNTAŞ, Study Director — Medipol University; Murat ATMACA, Study Chair — Medipol University; Sümeyye TUNÇ, Principal Investigator — Medipol University; Çağrı ÇAKICI, Study Chair — Medipol University; Türkan YİĞİTBAŞI, Study Chair — Medipol University
Locations (1):
- Sümeyye TUNÇ, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No